CLINICAL TRIAL: NCT00454350
Title: A Randomized , Open-Label, Cross-over, Pharmacokinetic Study of Doxercalciferol and Paricalcitol Following Multiple Intravenous Injections in Chronic Kidney Disease Subjects on Hemodialysis
Brief Title: A Phase 4 Pharmacokinetic Study of Hectorol Injection and Zemplar Injection in CKD Subjects on Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HECT00106
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Hectorol (doxercalciferol injection); Zemplar (paricalcitol injection)
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — 1 alpha-hydroxyergocalciferol; paricalcitol

INTERVENTIONS:
Drug: Hectorol (doxercalciferol injection)
Drug: Zemplar (Paricalcitol injection)

SUMMARY:
This study will measure serum levels of the active Vitamin D compound that circulates in hemodialysis subjects treated with either doxercalciferol injection (Hectorol®) or Zemplar® (paricalcitol injection).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be receiving hemodialysis three times per week for a minimum of three months.
* The subject must be receiving intravenous doxercalciferol or paricalcitol at each dialysis session (three times weekly) for a minimum of 12 weeks prior to Screening.
* At Screening Visit the subject's laboratory measurements must be within the following ranges: Serum iPTH measurement between 150-800 pg/mL; Corrected calcium measurement ≤ 10.5 mg/dL; Serum phosphorus measurement ≤ 7 mg/dL

Exclusion Criteria:

* Any ongoing use of over the counter or prescription vitamin D preparations except doxercalciferol or paricalcitol injection or multivitamins.
* History of heparin-induced thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Study | 44 hour interval

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Minneapolis, Minnesota, United States

REFERENCES:
- See also: US FDA Approved Full Prescribing Information for Hectorol® Injection — http://www.hectorol.com/docs/Hectorol%20Injection%20PI%20Text_2006-01.pdf